CLINICAL TRIAL: NCT00918996
Title: The Bladder Flap at Cesarean Delivery: Establishing Evidence for Practice
Brief Title: The Bladder Flap at Cesarean Section: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Methodius Tuuli, MD, MPH, Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRPO # 09-0173
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Cesarean Section
Keywords: Cesarean Section; Bladder Flap; Operating time

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Bladder Flap Group (Experimental): Uterine incision made 1 cm above the vesico-uterine reflection without incision and dissection of the bladder peritoneum.
  Interventions: Procedure: Omission of Bladder Flap Creation
- Bladder Flap Group (No Intervention): Standard cesarean section technique with incision and dissection of a bladder flap prior to uterine incision.

INTERVENTIONS:
Procedure: Omission of Bladder Flap Creation — Omission of bladder flap creation by making uterine incision 1 cm above the vesico-uterine reflection without incision and dissection of the bladder peritoneum.
  Other Names: No Flap
  Arms: No Bladder Flap Group

SUMMARY:
Cesarean section is now the most common major surgical procedure performed on women world wide. In the United States, approximately 1 in 4 deliveries is by this method. With the increasing numbers of cesarean sections, there is the need to utilized evidence based techniques to optimize outcomes and minimize complications.Creation of the bladder flap is an integral step of the standard cesarean section. The bladder flap is made by superficially incising and dissecting the peritoneal lining to separate the urinary bladder from the lower uterine segment. Started in the pre-antibiotic era, the rationale for the bladder flap was to enable the surgeon gain access to the lower uterine segment while minimizing injury to the bladder. Its subsequent closure was supposed to protect the peritoneal cavity from intrauterine infection. Since then, closure of the bladder flap has been demonstrated to be unnecessary and has been abandoned. The bladder flap however, continues to be performed without evidence of benefit.

Evidence on the role of the bladder flap in cesarean section is very limited. In emergent cesarean sections where rapid delivery is the goal, the bladder flap is commonly omitted. A simplified method of cesarean section (Pelosi-type) including omission of the bladder among other modifications has been shown to be safe and cost saving. The single randomized trial on omission of the bladder flap as the only modification suggests short term benefits including shorter operating times, reduced blood loss and decreased postoperative analgesic requirements. This study has been criticized for evaluating only short term outcomes and including only primary cesarean sections. The paucity of evidence for or against this commonly utilized technique in cesarean section is the rationale for this study.

The goal of this study is to employ a well designed randomized controlled clinical trial to evaluate the effects of omitting the bladder flap creation at cesarean section. We hypothesize that omission of the bladder flap in both primary and repeat cesarean sections will be associated with shorter operating time without a significant increase in intraoperative and postoperative complications.

DETAILED DESCRIPTION:
BACKGROUND

Cesarean section is the most common major surgical procedure in women world wide. In the United States almost 25% of deliveries are by cesarean section and the rate continues to rise [1]. In performing this procedure, it is imperative that evidence based techniques are utilized to optimize outcomes and minimize complications. Recently, the case has been made for simplifying the procedure by eliminating unnecessary and potentially harmful steps [2].

Rationale for the Bladder Flap Challenged: While the creation of the bladder flap has long been an integral part of the standard cesarean section, there is no evidence of benefit. Creation of the bladder flap at cesarean section dates back to the pre-antibiotic era of the 19th century. One rationale was to enable the surgeon gain access to the lower uterine segment while minimizing injury to the bladder [3]. While some older case reports suggested inadequate bladder flap reflection as a risk factor for bladder injury, it has not been collaborated [4]. On the contrary, several studies have identified difficulty encountered while developing the bladder flap as a risk factor for bladder injury at cesarean section [5, 6]. Although uncommon, creation of the bladder flap may also be associated with complications such as bladder flap hematoma and dysuria, sometimes requiring re-operation to drain the collection or release the bladder flap [7-11]. It has also been suggested that disruption of the autonomic innervations by creation of the bladder flap results in an increased incidence of urinary retention. In the long term, creation of the bladder flap may result in thick adhesions in the lower uterine segment that may lead to difficult subsequent cesarean delivery and bladder perforation [3].

Another rationale for the creation and subsequent closure of the bladder flap was to protect the peritoneal cavity from intrauterine infection. With the use of antibiotics, closure of the bladder flap has been demonstrated to be unnecessary and associated with increased morbidity including febrile morbidity, adhesions and upward dislocation of the urinary bladder [12, 13]. This evidence resulted in abandonment of closure of the bladder flap at cesarean section. Yet its creation has remained part of standard practice.

Limited Data on Role of Bladder Flap: Data on the role of the bladder flap in cesarean section is very limited. A simplified method of cesarean section (Pelosi-type) involving omission of the bladder among other modifications has been shown to be safe and cost saving [2]. Only one published study evaluated omission of the bladder flap as the only modification [14]. This single randomized trial compared omission of the bladder flap in 53 patients to the standard technique of cesarean section in 49 patients. The results showed significant short term benefits of omitting the bladder flap including a reduction in operating time, blood loss, postoperative pain and microhematuria.

The value of this European study is limited by the exclusion of repeat cesarean sections, lack of medium and long-term outcome measures such as adhesions as well as homogeneity of the study population. It has also been argued that the time saved from omitting the bladder flap (an average of 5 minutes) is not clinically significant [15]. On the other hand, 5 minutes saved for each of the 1 million cesarean sections performed annually in the United States will result in 1 million minutes (16667 hours, 694 days) of operating room time saved. Of note, this study was not designed to evaluate the effect of omitting the bladder flap on major bladder injuries. As the authors rightly argued, the low incidence of major bladder injuries at cesarean section (0.14-0.31%) means that a very large samples size (>40,000) would be required to demonstrate a difference [5, 16]. Such a study may never be done. The study was also limited to primary cesarean sections. The absence of data on omission of the bladder flap at repeat cesarean sections is particularly noteworthy. It is in these cases that adhesions in the lower uterine segment make creation of the bladder flap difficult and time consuming, with the potential for complications.

The only other report on the effects of omitting the bladder flap at cesarean section is a West African case series of 142 patients [17]. That data is of little value, given the absence of a comparison group and the unique study setting.

Evidence needed for Practice: From the above, it appears that the wide spread use of the bladder flap at cesarean section is based more on anecdotal evidence and clinical impression than scientific evidence [3]. At present, it remains to be established if there is any advantage in dissecting the bladder from the lower uterine segment during cesarean section. The paucity of evidence for this commonly utilized technique in cesarean section calls for a well designed randomized trial to provide the much needed evidence to inform clinic practice. With the increasing numbers of cesarean deliveries, eliminating unnecessary and potentially harmful steps will reduce morbidity, improve outcomes and save costs.

RESEARCH OBJECTIVES

The goal of this study is to employ a well designed randomized controlled clinical trial to evaluate the effects of omitting the bladder flap creation at cesarean section. We hypothesize that omission of the bladder flap in both primary and repeat cesarean sections will be associated with shorter operating time without a significant increase in intraoperative and postoperative complications. Specifically, we propose:

Aim 1: To evaluate short term effects of omitting the bladder flap including duration of surgery, blood loss, hematuria and immediate postoperative pain;

Aim 2: To evaluate medium term effects of omitting the bladder flap such as persistent hematuria, dysuria, and ongoing requirement for pain control and

Aim 3: To evaluate long term effects of omitting the bladder flap including adhesions and duration of a subsequent cesarean section.

STUDY DESIGN AND METHODS

Study Design: This will be a randomized controlled trial comparing the effects of omission of the bladder flap to the standard cesarean section technique. Enrolled patients will be stratified into primary and repeat cesarean sections and then randomized by a computer based program into 'bladder flap' and 'no bladder flap' groups.

Recruitment: All eligible patients who are scheduled for cesarean sections from the Barnes Jewish and Center for Advanced Medicine OB/GYN clinics will be approached for consent to participate in the study. Patients will be given study information and the consent form to review at home. For unscheduled patients, consent will be sought once the decision has been made to perform a cesarean section. This will be limited to non-emergent indications, where consent can be obtained without interfering with patient care.

Procedures: Before entering the operating room, the surgeon will open a sealed envelope containing the randomization number and the patient's allocation. The technique for cesarean section will be similar in each group, except for the omission or creation of the bladder flap. In the 'no bladder flap' group, a low-transverse uterine incision will be performed about 1cm above the vesicouterine peritoneal fold, without dissection and formation of a bladder flap [14]. Patients will undergo the procedure based on their allocation unless intraoperative findings as determined by the surgeon make the alternative procedure medically indicated. Demographic (e.g. age, race, socioeconomic status), obstetric (e.g. parity, gestational age, indication for cesarean section, cervical dilation at time of cesarean section, presence of chorioamnionitis, surgical complications) and neonatal (e.g. birth weight, Apgar score, cord pH) data will be abstracted from the patients chart.

Follow up Study: We plan a follow up to this study aimed at evaluating long term effects of omitting the bladder flap. All enrolled patients who subsequently undergo a repeat cesarean section in our facility within 5 years will be assessed for the duration of the subsequent surgery and the amount of intraperitoneal adhesions. A previously published adhesion score system which includes location and degree of adhesions will be used [18]. The surgeon in the repeat cesarean section will be blinded to the initial allocation of the patient.

Data Analysis: Analysis of the primary outcome and most other analyses will be performed separately within the primary and the repeat cesarean section groups as well as in the combined study population. Analyses will be based on intent to treat. Surgical time and secondary outcome such as blood loss will be compared across groups using unpaired t-tests. However, if blood loss is identified to be a skewed variable, it is possible that we will use Wilcoxon's test or alternatively, use the t-test following a log transformation of the data. If a significant variation is noted in individual surgeons' operating times, further analysis will adjust for this using the surgeon's operating time index, defined as operating time / mean surgeon's operating time. These analyses will be supplemented with multiple regression analyses that adjust for covariates that include the age of the mother, gestational age, indication for the cesarean section, and cervical dilation at the time of the surgery that are identified to be potential confounding variables. Secondary outcomes such as hematuria and whether pain medication is still required at 2-4 weeks will be analyzed using chi square tests, with logistic regression being employed to assess significance after adjusting for the relevant covariates listed above. A final set of linear and logistic regression analyses will include both primary and repeat cesarean sections and will evaluate the interaction between the use of the bladder flap and whether the surgery type is primary or repeat to see if the impact of the bladder flap is different in one subgroup as compared to the other. Analyses will be performed using Stata version 10 (Stata Corp., College Station, TX).

Sample size considerations: Since the goal of this study is to evaluate the impact of the bladder flap separately in primary and repeat cesarean section patients, we provide separate power computations for these two groups. Based on a mean duration of 45 minutes(SD 10minutes)for primary cesareans and an anticipated saving of 5 minutes from omitting the bladder flap, our target sample size will be 64 primary cesarean sections per group, to yield a statistical power of 0.8 for a two-sided test at the 0.05 level of significance. For the repeat cesarean sections we anticipate a larger time saving due to the impact of scar tissue. However, to be conservative, we assume a 5 minute time saving in this group as well. We incorporate an interim efficacy analysis into this group and, using the Obrien-Fleming stopping rule to adjust for type I error, we base our power computations on a nominal p-value of 0.047. With this nominal pvalue, the sample size requirement is 65 per group for a power of 0.8 to detect a 5-minute operative time difference for a two-sided test at the 0.05 level of significance. Thus, a total of 258 patients will be recruited (64 x 2 + 65 x 2).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-emergent primary and repeat cesarean sections at or greater than 32 weeks gestation at Barnes Jewish Hospital during the study period.

Exclusion Criteria:

* Emergent cesarean sections, planned vertical uterine incision, previous abdominal surgeries (besides prior cesarean sections), sedation and inability to obtain consent.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Total operating time (from skin incision to closure of the skin). | Intraoperative

SECONDARY OUTCOMES:
Skin incision to delivery time, skin incision to fascial closure time, blood loss, hematuria, dysuria, urinary retention, febrile morbidity, use of analgesics, hospital days, wound infection, endomyometritis, neonatal outcomes, and readmissions. | On first postoperative day and at 2-4 week postoperative visit

CONTACTS AND LOCATIONS:
Overall Officials: George A. Macones, MD, MSCE, Principal Investigator — Washington University School of Medicine; Methodius G. Tuuli, M.D., M.P.H., Principal Investigator — Washington University School of Medicine; Anthony Odibo, MD, MSCE, Principal Investigator — Washington University School of Medicine; Patricia Fogertey, BSN, MSN, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Hamilton BE, Martin JA, Ventura SJ. Births: preliminary data for 2005. Natl Vital Stat Rep. 2006 Dec 28;55(11):1-18. PMID 17432301
- [Background] Wood RM, Simon H, Oz AU. Pelosi-type vs. traditional cesarean delivery. A prospective comparison. J Reprod Med. 1999 Sep;44(9):788-95. PMID 10509303
- [Background] Pelosi MA 2nd, Pelosi MA 3rd. Risk factors for bladder injury during cesarean delivery. Obstet Gynecol. 2005 Apr;105(4):900; author reply 901. doi: 10.1097/01.AOG.0000158756.29999.0a. No abstract available. PMID 15802429
- [Background] Faricy PO, Augspurger RR, Kaufman JM. Bladder injuries associated with cesarean section. J Urol. 1978 Dec;120(6):762-3. doi: 10.1016/s0022-5347(17)57354-1. PMID 731822
- [Background] Eisenkop SM, Richman R, Platt LD, Paul RH. Urinary tract injury during cesarean section. Obstet Gynecol. 1982 Nov;60(5):591-6. PMID 7145252
- [Background] Rahman MS, Gasem T, Al Suleiman SA, Al Jama FE, Burshaid S, Rahman J. Bladder injuries during cesarean section in a University Hospital: a 25-year review. Arch Gynecol Obstet. 2009 Mar;279(3):349-52. doi: 10.1007/s00404-008-0733-1. Epub 2008 Jul 22. PMID 18648828
- [Background] Acholonu F, Minkoff H, Delke I. Percutaneous drainage of fluid collections in the bladder flap of febrile post-cesarean-section patients. A report of seven cases. J Reprod Med. 1987 Feb;32(2):140-3. PMID 3560077
- [Background] Baker ME, Bowie JD, Killam AP. Sonography of post-cesarean-section bladder-flap hematoma. AJR Am J Roentgenol. 1985 Apr;144(4):757-9. doi: 10.2214/ajr.144.4.757. PMID 3883710
- [Background] Jozwik M, Jozwik M, Lotocki W, Mironczuk J. Dysuria due to bladder distortion after repeat cesarean section. Gynecol Obstet Invest. 1998;45(4):279-80. doi: 10.1159/000009985. PMID 9623798
- [Background] Malvasi A, Tinelli A, Tinelli R, Rahimi S, Resta L, Tinelli FG. The post-cesarean section symptomatic bladder flap hematoma: a modern reappraisal. J Matern Fetal Neonatal Med. 2007 Oct;20(10):709-14. doi: 10.1080/01674820701450573. PMID 17763270
- [Background] Winsett MZ, Fagan CJ, Bedi DG. Sonographic demonstration of bladder-flap hematoma. J Ultrasound Med. 1986 Sep;5(9):483-7. doi: 10.7863/jum.1986.5.9.483. PMID 3531540
- [Background] Woyton J, Florjanski J, Zimmer M. [Nonclosure of the visceral peritoneum during Cesarean sections]. Ginekol Pol. 2000 Oct;71(10):1250-4. Polish. PMID 11143933
- [Background] Nagele F, Karas H, Spitzer D, Staudach A, Karasegh S, Beck A, Husslein P. Closure or nonclosure of the visceral peritoneum at cesarean delivery. Am J Obstet Gynecol. 1996 Apr;174(4):1366-70. doi: 10.1016/s0002-9378(96)70686-5. PMID 8623871
- [Background] Hohlagschwandtner M, Ruecklinger E, Husslein P, Joura EA. Is the formation of a bladder flap at cesarean necessary? A randomized trial. Obstet Gynecol. 2001 Dec;98(6):1089-92. doi: 10.1016/s0029-7844(01)01570-8. PMID 11755558
- [Background] Honig J. Is the formation of a bladder flap at cesarean necessary? A randomized trial. Obstet Gynecol. 2002 Apr;99(4):677; author reply 677-8. doi: 10.1016/s0029-7844(02)01925-7. No abstract available. PMID 12039137
- [Background] Rajasekar D, Hall M. Urinary tract injuries during obstetric intervention. Br J Obstet Gynaecol. 1997 Jun;104(6):731-4. doi: 10.1111/j.1471-0528.1997.tb11986.x. PMID 9197879
- [Background] Chigbu CO, Ezeome IV, Iloabachie GC. Non-formation of bladder flap at cesarean section. Int J Gynaecol Obstet. 2006 Dec;95(3):284-5. doi: 10.1016/j.ijgo.2006.08.010. Epub 2006 Oct 23. No abstract available. PMID 17056044
- [Background] Lyell DJ, Caughey AB, Hu E, Daniels K. Peritoneal closure at primary cesarean delivery and adhesions. Obstet Gynecol. 2005 Aug;106(2):275-80. doi: 10.1097/01.AOG.0000171120.81732.4c. PMID 16055575
- [Derived] Tuuli MG, Odibo AO, Fogertey P, Roehl K, Stamilio D, Macones GA. Utility of the bladder flap at cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2012 Apr;119(4):815-21. doi: 10.1097/AOG.0b013e31824c0e12. PMID 22395144